CLINICAL TRIAL: NCT04412915
Title: Correlation Between Early Induction of Labor and Cesarean Delivery in Low-risk Nulliparous Women
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 109050-F
Record Dates: First submitted 2020-05-31; First posted 2020-06-02 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-12

CONDITIONS: Low Risk Pregnancy
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Labor induction — Labor induction with oxytocin or prostagladin

SUMMARY:
To elucidate whether induction of labor in primiparas with low-risk pregnancies at 38 + 0 to 40 + 6 gestational weeks will increase the cesarean rate, compared with those receiving labor induction at more than 41+0 gestational weeks.

DETAILED DESCRIPTION:
Medical records of all consecutive primiparas with low-risk pregnancy from January 1, 2014 to August 31, 2019 were reviewed to explore the correlation between early induction of labor and caesarean birth after 38 + 0 weeks. The hypothesis of the study is that induction of labor in primiparas with low-risk pregnancies at 38 + 0 to 40 + 6 gestational weeks will increase the cesarean rate, compared with those receiving labor induction at more than 41+0 gestational weeks.

ELIGIBILITY:
Inclusion Criteria:

* After 38 + 0 weeks of gestation
* low-risk pregnant primiparas
* singleton
* nulliparous
* > 20 years old

Exclusion Criteria:

* Premature rupture of membranes

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — primiparas
Study Population: Medical records of all consecutive primiparas with low-risk pregnancy from January 1, 2014 to August 31, 2019
Sampling Method: Non-Probability Sample
Enrollment: 2125 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Cesarean rate rate | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan